CLINICAL TRIAL: NCT06580717
Title: ENavogliflozin DElivering Alleviation of Ventricular Diastolic Dysfunction in nonObstRuctive Hypertrophic CardioMyopathy: a Prospective, Multicenter, Randomized, Double-blind, Placebo-controlled Study (ENDEAVOR-HCM)
Brief Title: ENavogliflozin DElivering Alleviation of Ventricular Diastolic Dysfunction in nonObstRuctive Hypertrophic CardioMyopathy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2024-0089
Record Dates: First submitted 2024-03-25; First posted 2024-08-30 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Nonobstructive Hypertrophic Cardiomyopathy
Keywords: non-obstructive; SGLT2; hypertrophic cardiomyopathy; HCM; ENDEAVOR-HCM; ertugliflozin
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — Enavogliflozin

STUDY DESIGN:
Who Masked: Participant
Masking Description: Researchers, research coordinators, and subjects are all blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enavogliflozin 0.3mg (Experimental): Patients who are eligible for all of the criteria and who do not qualify as exclusion criteria should be enrolled in the study and randomly enrolled in a 1: 1 dose of enavogliflozin 0.3 mg once daily or placebo.
  Interventions: Drug: enavogliflozin 0.3mg
- Enavogliflozin placebo (Placebo Comparator): Patients who are eligible for all of the criteria and who do not qualify as exclusion criteria should be enrolled in the study and randomly enrolled in a 1: 1 dose of enavogliflozin 0.3 mg once daily or placebo.
  Interventions: Drug: enavogliflozin Placebo

INTERVENTIONS:
Drug: enavogliflozin 0.3mg — Enavogliflozin 0.3mg, 1 tablet once a day, is prescribed for a period of 24 weeks.
  Patients who are eligible for all of the criteria and who do not qualify as exclusion criteria should be enrolled in the study and randomly enrolled in a 1: 1 dose of enavogliflozin 0.3 mg once daily or placebo.
  Arms: Enavogliflozin 0.3mg
Drug: enavogliflozin Placebo — A placebo pill identical to enavogliflozin, 1 tablet once a day, is prescribed for a period of 24 weeks.
  Patients who are eligible for all of the criteria and who do not qualify as exclusion criteria should be enrolled in the study and randomly enrolled in a 1: 1 dose of enavogliflozin 0.3 mg once daily or placebo.
  Arms: Enavogliflozin placebo

SUMMARY:
The primary objective of this study is to investigate the effect of enavogliflozin, an Sodium-glucose transporter 2 (SGLT2) inhibitor, compared with placebo on left ventricular diastolic function in patients with nonobstructive hypertrophic cardiomyopathy. The secondary objective of this study is to investigate the effect of enavogliflozin on exercise capacity, symptoms, serum biomarkers, and arrhythmic burden in patients with nonobstructive hypertrophic cardiomyopathy.

DETAILED DESCRIPTION:
Most of the medication used in HCM(hypertrophic cardiomyopathy) targets dynamic left ventricular obstruction and hypercontractility. Guidelines recommend that beta-blockers and calcum channels can also be used to lower heart rate and improve diastolic function in symptomatic nonobstructive HCM(hypertrophic cardiomyopathy), and that diuretics may be considered next, but there is a paucity of evidence supporting these recommendations. Left ventricular diastolic dysfunction is the main pathophysiological mechanism in nonobstructive HCM. SGLT2(Sodium-glucose transporter 2) inhibitors have been shown to reduce heart failure events and mortality in patients with heart failure with preserved ejection fraction, and have also been reported to improve left ventricular diastolic function. This study will investigate the efficacy and safety of enavogliflozin, an SGLT2(Sodium-glucose transporter 2) inhibitor, compared with placebo in patients with nonobstructive hypertrophic cardiomyopathy, over a period of 6 months.

Patients with hypertrophic cardiomyopathy and without evidence of dynamic left ventricular outflow tract obstruction at resting or on provocation by Valsalva maneuver or exercise will be enrolled. Participants will be randomly assigned to the enavogliflozin 0.3mg group and the placebo group in a 1:1 ratio and will continue the medication for 24 weeks. Changes in left ventricular diastolic reserve assessed by diastolic stress echocardiography will be compared between the treatment groups at 24 weeks. Changes in other parameters of diastolic function and exercise capacity will be assessed by diastolic stress echocardiography and compared between the treatment groups. Symptom status, serum biomarker levels, and arrhythmic burden on 24 hour ambulatory electrocardiogram will also be compared between the treatment groups. Post-trial follow-up will be performed at 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. A patient who understands the research protocol and fills out a consent form
2. Adults over 19 years of age and under 80 years of age
3. Non-diabetic or type 2 diabetic patients (HbA1c 6.5-10.5%)
4. Patients with non-obstructive hypertrophic cardiomyopathy who do not show significant dynamic left ventricular outflow tract obstruction at rest or during Valsalva maneuver or exercise stress on echocardiography within 3 months of the screening visit.

   * Non-obstructive hypertrophic cardiomyopathy: corresponds to maximum left ventricular outflow tract pressure gradient <30mmHg.
   * Maximum left ventricular wall thickness ≥15mm if there is no family history of hypertrophic cardiomyopathy, or maximum left ventricular wall thickness ≥13mm if there is a family history of hypertrophic cardiomyopathy or positive for related genetic mutation.
5. For hypertrophic cardiomyopathy, existing beta blockers, calcium channel blockers, diuretics and Renin-angiotension-system(RAS) blockers (beta-blocker, non-dihydropyridine Calcium Cannel Blocker, loop diuretics, thiazide and thiazide-like diuretics, mineralocorticoid receptor antagonist, angiotensin converting enzyme inhibitor/angiotensin) For patients using receptor blocker/angiotensin receptor neprilysin inhibitor), the drug dose was stable for 2 weeks before screening and no change in dose is expected throughout the study period.
6. Women of childbearing age who agree to use contraception (hormones, intrauterine device, tubal ligation, spouse's vasectomy, etc.) for 30 days from the time of screening, during the clinical trial period, and after taking the clinical trial drug.
7. New York Heart Association (NYHA) Class 1~3

Exclusion Criteria:

1. History of hypersensitivity to clinical trial drugs
2. If you are currently taking Sodium-glucose transporter 2 (SGLT2) inhibitors or within 4 weeks

   - For diabetic patients, any type of hypoglycemic agent other than Sodium-glucose transporter 2 (SGLT2) inhibitors can be used.
3. Patients who cannot undergo diastolic stress echocardiography
4. Patients on dialysis or with chronic renal failure with an estimated glomerular filtration rate <30 mL/min/1.73m2
5. Patients with Cardiac implantable electronic device (CIED)
6. Currently pregnant or lactating
7. ASpartate Transaminase(AST) or ALanine Transaminase(ALT) value more than 3 times the upper limit of normal during liver function test, history of hepatic coma, history of esophageal varices, history of porto-caval anastomosis.
8. Uncontrolled hypertension (SBP≥180mmHg or DBP≥110mmHg) or severe hypotension (SBP<90mmHg)
9. Severe aortic or mitral stenosis with the possibility of surgery during the clinical trial period
10. Those waiting for a heart transplant or those who have received a heart transplant
11. Persons with diseases that need to be differentiated from heart failure symptoms at the investigator's discretion, such as severe anemia (hemoglobin <7 g/dL), uncontrolled arrhythmia, severe lung disease, etc.
12. If you have cancer undergoing chemotherapy/radiation/surgical treatment or if your life expectancy is expected to be less than 1 year.
13. Untreated alcohol or drug abuse
14. If you are participating in the administration of another clinical trial drug or clinical trial device test, or have completed participation for less than 30 days.
15. Patients with type 1 diabetes or diabetic ketoacidosis
16. New York Heart Association (NYHA) class 4

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in left ventricular diastolic reserve (Δe') assessed by diastolic stress echocardiography | 24 weeks, 52 weeks
  This variable will be assessed by diastolic stress echocardiography and compared to baseline values at 24 weeks (end of study) This variable will be assessed by diastolic stress echocardiography and compared to baseline values at 52 weeks (post-trial 24 weeks).
  This variable will be assessed by diastolic stress echocardiography and compared to 24 weeks (end of study) values at 52 weeks (post-trial 24 weeks).

SECONDARY OUTCOMES:
Comparison of Diastolic Stress Echocardiography Parameters | 24 weeks, 52 weeks
  Change from enrollment to end of study in e' (cm/sec) at 52 weeks
  Change from enrollment to end of study in E (m/sec) at 52 weeks
  Change from enrollment to end of study in E to e' ratio at 52 weeks
  Change from enrollment to end of study in pulmonary artery systolic pressure (mmHg) at 52 weeks
  Change from enrollment to end of study in global longitudinal left ventricular strain (%) at 52 weeks
  Change from enrollment to end of study in left atrial reservoir strain (%) at 52 weeks
Comparison of Cardiopulmonary Exercise Testing Parameters | 24 weeks, 52 weeks
  Change from enrollment to end of study in peak oxygen consumption (VO2max) (ml/kg/min) at 52 weeks
  Change from enrollment to end of study in VE to VCO2 slope (ratio) at 52 weeks
  Change from enrollment to end of study in ventilatory anaerobic threshold (VAT) (ml/kg/min) at 52 weeks
  Change from enrollment to end of study in metabolic equivalents (METs) at 52 weeks
  Change from enrollment to end of study in exercise time (min) at 52 weeks
Comparison of Blood Biomarkers | 24 weeks, 52 weeks
  Change from enrollment to end of study in NT-proBNP levels (pg/mL) at 52 weeks.
  Change from enrollment to end of study in Troponin T levels (ng/mL) at 52 weeks.
Comparison of Symptom Survey | 24 weeks, 52 weeks
  Change from enrollment to end of study in New York Heart Association (NYHA) Functional Class (Functional class I, II, III, IV) at 52 weeks
  Change from enrollment to end of study in Kansas City Cardiomyopathy Questionnaire (KCCQ) Overall Summary Score (0 to 100, with higher scores indicating better health.) at 52 weeks
Comparison of Arrhythmic Burden on 24-Hour Ambulatory Electrocardiogram | 24 weeks, 52 weeks
  Change from enrollment to end of study in Atrial Premature Contractions(APC) burden at 52 weeks
  Change from enrollment to end of study in Ventricular Premature Contractions(VPC) burden at 52 weeks
  Change from enrollment to end of study in APC to VPC burden ratio (%) at 52 weeks
  Change from enrollment to end of study in Standard Deviation of Normal Sinus R-R Intervals (SDNN) (ms) at 52 weeks.
  Change from enrollment to end of study in root mean square of the mean of the squared differences of two consecutive R-R intervals (rMSSD) (ms) at 52 weeks.
  Change from enrollment to end of study in Low Frequency(LF) to High Frequency(HF) ratio at 52 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Jiwon Seo, MD, Principal Investigator — Gangnam Severance Hospital; Jang-Won Son, MD, Principal Investigator — Yeungnam University Hospital; In-Cheol Kim, MD, Principal Investigator — Keimyung University Dongsan Medical Center
Locations (1):
- Division of Cardiology, Yonsei Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No